CLINICAL TRIAL: NCT02877758
Title: Investigation of a Novel Cosmeceutical to Reduce the Visible Signs of Cutaneous Aging - A Randomized Controlled Double Blind Study
Brief Title: Investigation of a Novel Cosmeceutical to Reduce the Visible Signs of Cutaneous Aging
Acronym: REDUCEAGE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tomorrowlabs GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMRW-CTa
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Aging
Keywords: cutaneous aging; skin rejuvenation; wrinkles
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Tomorrowlabs cosmeceutical formulation is applied to the face of the subjects twice daily for 3 consecutive months.
  Interventions: Other: Tomorrowlabs cosmeceutical formulation
- Control (Sham Comparator): Tomorrowlabs cosmeceutical formulation without the active ingredient is applied to the face of the subjects twice daily for 3 consecutive months.
  Interventions: Other: Sham cosmeceutical formulation

INTERVENTIONS:
Other: Tomorrowlabs cosmeceutical formulation
  Other Names: HSF Cellular Age Reversal and Repair; HSF Day Catalyst
  Arms: Experimental
Other: Sham cosmeceutical formulation
  Arms: Control

SUMMARY:
Tomorrowlabs has developed a revolutionary cosmeceutical formulation to rejuvenate aging skin. Tomorrowlabs is conducting this research to study whether this cosmeceutical can reduce the visible signs of cutaneous aging.

DETAILED DESCRIPTION:
It is proposed to study a cosmeceutical formulation designed to reduce the visible signs of cutaneous aging. It is expected that daily application of the formulation may minimize wrinkles and fine lines of the face.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who desire to improve their appearance by reducing the visible signs of cutaneous aging in the face

Exclusion Criteria:

* Subjects who have undergone facial plastic surgery or aesthetic dermatology treatments to the face (such as fillers and neuromodulators) in the past 6 months
* Subjects with a history of collagen vascular disease, cutis laxa, connective tissue disease, psoriasis, or lupus.
* Subjects diagnosed with scleroderma.
* Subjects with a body mass index (BMI) > 30.
* Subjects taking steroid therapy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Validated Assessment Scales for Age-related Changes of the Face | 3 months
  A reliable tool for valid and reproducible assessment of the aging process in various face areas will be employed by our independent panel of assessors to scale the primary outcome. (1-3)

SECONDARY OUTCOMES:
Skin quality assessment | 3 months
  The skin scope uses black light and magnification to show variety of skin imperfections that are undetectable with the naked eye such as dry and thin skin
Subject Satisfaction With the Results | 3 months
  Self assessment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Wenny, MD, Principal Investigator — JKU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Narins RS, Carruthers J, Flynn TC, Geister TL, Gortelmeyer R, Hardas B, Himmrich S, Jones D, Kerscher M, de Maio M, Mohrmann C, Pooth R, Rzany B, Sattler G, Buchner L, Benter U, Breitscheidel L, Carruthers A. Validated assessment scales for the lower face. Dermatol Surg. 2012 Feb;38(2 Spec No.):333-42. doi: 10.1111/j.1524-4725.2011.02247.x. PMID 22316189
- [Background] Carruthers J, Flynn TC, Geister TL, Gortelmeyer R, Hardas B, Himmrich S, Jones D, Kerscher M, de Maio M, Mohrmann C, Narins RS, Pooth R, Rzany B, Sattler G, Buchner L, Benter U, Breitscheidel L, Carruthers A. Validated assessment scales for the mid face. Dermatol Surg. 2012 Feb;38(2 Spec No.):320-32. doi: 10.1111/j.1524-4725.2011.02251.x. PMID 22316188
- [Background] Flynn TC, Carruthers A, Carruthers J, Geister TL, Gortelmeyer R, Hardas B, Himmrich S, Kerscher M, de Maio M, Mohrmann C, Narins RS, Pooth R, Rzany B, Sattler G, Buchner L, Benter U, Fey C, Jones D. Validated assessment scales for the upper face. Dermatol Surg. 2012 Feb;38(2 Spec No.):309-19. doi: 10.1111/j.1524-4725.2011.02248.x. PMID 22316187